CLINICAL TRIAL: NCT05017324
Title: Sequencing Mycobacteria and Algorithm-determined Resistant Tuberculosis Treatment Trial
Acronym: SMARTT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiteit Antwerpen (Other)
Collaborators: Aurum Institute (Other); University of Stellenbosch (Other); University of the Free State (Unknown); Free State Department of Health (Unknown)
Responsible Party: Principal Investigator, Annelies Van Rie, Professor, Universiteit Antwerpen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AUR1-11-248; T001018N (Other Grant/Funding Number: TBM FWO); 2020-004084-10 (EudraCT Number)
Record Dates: First submitted 2021-04-22; First posted 2021-08-23 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Rifampicin Resistant Tuberculosis; Drug-resistant Tuberculosis; Multidrug Resistant Tuberculosis; Pulmonary Tuberculoses
Keywords: Whole Genome Sequencing; Drug Resistant Tuberculosis
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant; Tuberculosis, Pulmonary

STUDY DESIGN:
Intervention Model Description: Randomized Controled Phase 4 pragmatic single blinded medical device trial.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WGS DST strategy (Experimental): WGS DST strategy for diagnosing the TB drug resistance profile and an individualised RR-TB treatment recommendation
  Interventions: Device: WGS DST strategy
- Standard of Care (No Intervention): Standard of care diagnosis of the drug resistance profile and individualised treatment

INTERVENTIONS:
Device: WGS DST strategy — WGS DST strategy for diagnosing the TB drug resistance profile and an algorithm-determined individualised RR-TB treatment recommendation
  Arms: WGS DST strategy

SUMMARY:
The primary aim of this pragmatic trial is to determine the effectiveness of a Whole Genome Sequencing (WGS) Drug Sensitivity Testing (DST) strategy to guide individualised treatment of rifampicin resistant tuberculosis (RR-TB) patients.

The primary objective is to determine the effectiveness of this WGS DST strategy in patients diagnosed with RR-TB. We will additionally perform an exploratory health economics evaluation of both arms, and will determine the feasibility of the WGS DST strategy.

DETAILED DESCRIPTION:
The trial will be a single blinded randomised controlled, pragmatic, medical device trial evaluating a Whole Genome Sequencing (WGS) Drug Sensitivity Testing (DST) strategy to guide individualised treatment of rifampicin resistant tuberculosis (RR-TB) patients. A total of 248 patients diagnosed with RR-TB in the South African Free State province will by randomised to one of two trial arms. 124 patients will be assigned to the intervention arm, consisting of a WGS DST strategy for diagnosing drug resistance profile and an algorithm-determined individualised RR-TB treatment recommendation. 124 patients will be assigned to the control arm where the diagnosis of Mtb drug resistance and individualisation of RR-TB treatment will happen according to the Standard of Care (SOC) procedures.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with RR-TB
* Diagnosed with pulmonary TB (PTB) or PTB plus extra-pulmonary TB (EPTB)
* ≥18 years of age
* Able to sign informed consent
* Not on TB treatment at time of enrolment

Exclusion Criteria:

* Patients diagnosed EPTB without pulmonary involvement
* Patients with TB Meningitis or TB of the bone.
* Has any condition that, in the opinion of the investigator or physician, would preclude provision of informed consent, make participation in the study unsafe, complicate interpretation of study outcome data, interfere with achieving the study objectives or compromise patient safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2021-09-21 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
The Effectiveness of a WGS DST strategy for individualisation of RR-TB treatment | Day 0 to month 6 (6 months)
  The effectiveness will be determined by the rate of change in time to positivity (TTP) over 6 months in the Mycobacterial Growth Indicator Tuber (MGIT) system [time from: Day 0 to Week 24].
  The effectiveness of the WGS DST strategy will be determined by the rate of change in TTP in liquid media MGIT cultures of sputum samples collected during the first 6 months of treatment. The TTP will be used to determine the change in mycobacterial load using a non-linear mixed effect time-to-event model that provides a longitudinal representation of mycobacterial load (measured as TTP in MGIT) at weeks 2, 3, 4, 5, 6, 7, 8, 12, 16, 20 and 24

SECONDARY OUTCOMES:
Health economic evaluation of a WGS DST strategy for individualization of RR-TB treatment | Start of treatment to end of treatment (which may vary from 6 months to over 11 months)
  The difference in total cost over the entire treatment period from a patients and health system perspective between a WGS strategy and SOC strategy will be assessed by comparing costing data collected at month 1 of treatment, month 6 of treatment and at the end of treatment.
Impact of WGS strategy for individualisation of RR-TB treatment on Health related Quality of Life (HRQOL) | Start of treatment to end of treatment (which may vary from 6 months to over 11 months)
  The difference in changes in health relates quality fo life will be assessed by comparing the change in HRQOL over time between patients randomised to the WGS and SOC strategies for individualisation of RR-TB treatment, using results of the EQ-5D-5L questionnaire collected at baseline, month 1, 2, 3, 4, 5, 6 and end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Gavin Churchyard, PhD, MD, Principal Investigator — Aurum Institute; Annelies Van Rie, PhD, MD, Principal Investigator — Universiteit Antwerpen; Rob M Warren, PhD, Principal Investigator — Stellenbosch University, MRC; Salome Charalambous, PhD, Principal Investigator — Aurum Institute
Locations (1):
- Free State Department of Health Clinics, Bloemfontein, Free State, South Africa

IPD SHARING:
Plan to Share IPD: Yes
The analysable individual patient data (IPD) will be made available, including WGS data (to be published on the European Nucleotide Archive (ENA)) and de-identified clinical and demographic IPD. This ensures an adit trial for summary results reporting, enables re-analyses of trial data and the possibility for combining the data with others for novel investigations.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From publication of the results of the primary up to 5 years thereafter
Access Criteria: WGS: available on European Nucleotide Archive (ENA) Other data: access will be provided to researchers who have obtained Institutional Review Board (IRB) approval for analyses

REFERENCES:
- [Derived] Van Rie A, De Vos E, Costa E, Verboven L, Ndebele F, Heupink TH, Abrams S; SMARTT team; Fanampe B, Van der Spoel Van Dyk A, Charalambous S, Churchyard G, Warren R. Sequencing Mycobacteria and Algorithm-determined Resistant Tuberculosis Treatment (SMARTT): a study protocol for a phase IV pragmatic randomized controlled patient management strategy trial. Trials. 2022 Oct 8;23(1):864. doi: 10.1186/s13063-022-06793-w. PMID 36209235